CLINICAL TRIAL: NCT04059536
Title: Performance and Safety of the Roxwood CenterCross™ CenterCross™ Ultra, CenterCross™ Ultra LV and MultiCross™ Catheters and MicroCross™ MicroCatheter in Native Coronary and Peripheral Arteries With a Stenotic Lesion or Chronic Total Occlusion (CTO)
Brief Title: Registry Study to Evaluate the Performance and Safety of Roxwood Medical Catheters in Arteries of Participants With a Stenotic Lesion or Chronic Total Occlusion (CTO)
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor decision
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: EKOS Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: BTG-007927-01
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Chronic Total Occlusion; Atherosclerosis; Coronary Artery Disease; Peripheral Artery Disease
Keywords: Stenotic Lesions
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease; Peripheral Arterial Disease | interventions — Aspirin; Heparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Roxwood Anchoring Catheters: Participants will be treated for an index procedure using Roxwood Medical device(s) as prescribed by the Investigator SOC on Day 0. All devices will be used in accordance with the Instructions for Use (IFU). Participants are to be administered SOC acetylsalicylic acid (ASA) and/or anti-platelet medications orally per physician discretion prior to the index procedure. Administration of an intravenous injection of heparin during the index procedure will also be at the discretion of the Investigator per Institutional SOC.
  Interventions: Device: Roxwood Anchoring Catheters; Drug: Acetylsalicylic Acid; Drug: Heparin

INTERVENTIONS:
Device: Roxwood Anchoring Catheters — Anchoring catheters
  Other Names: Roxwood CenterCross™ Catheter - 125 centimeters (cm) working length; CenterCross™ ULTRA Catheter - 125 cm working length; CenterCross™ ULTRA LV Catheter - 100 cm working length; MultiCross™ Catheter - 135 cm working length; MicroCross™ 14 Microcatheter- 135 cm working length; MicroCross™ 14 Microcatheter - 155 cm working length; MicroCross™ 14ES Extra Support Microcatheter - 135 cm working length; MicroCross™ 18 Microcatheter - 90 cm working length; MicroCross™ 18 Microcatheter - 135 cm working length; MicroCross™ 18 Microcatheter - 155 cm working length
Drug: Acetylsalicylic Acid — Oral Tablet
  Other Names: Aspirin
Drug: Heparin — Intravenous Injection

SUMMARY:
The purpose of this registry study is to gather real world standard of care (SOC) data on the safety and performance on the Roxwood Medical catheter devices in the treatment of stenotic lesions and CTO.

DETAILED DESCRIPTION:
The Roxwood Anchoring Catheters are a group of artery catheters used in participants undergoing interventional procedures. These anchoring catheters are support catheters used in conjunction with guidewires to access discrete regions of the coronary and peripheral vasculature. They may be used to facilitate placement and exchange of guidewires and/or other interventional devices beyond stenotic lesions, including CTOs. The goal of this registry study is to collect prospective observational data on the performance of the Roxwood CenterCross™, CenterCross™ Ultra, CenterCross™ Ultra LV, MultiCross™, and MicroCross™ 14, 14ES and 18 MicroCatheter devices through 24 hours and the safety of the devices through 30 days in native coronary and peripheral arteries with a stenotic lesion or CTO. Additionally, the catheters will be evaluated for the ability to facilitate a guidewire successfully penetrating the proximal cap of the stenotic lesion or CTO and the infusion of saline and contrast agents as confirmed by angiography.

Of the 100 intended participants to be treated, it is anticipated that at least 50 participants will be enrolled and treated using the Roxwood MicroCross™ 14, 14ES and/or 18 MicroCatheter and 50 participants will be enrolled and treated using the CenterCross™, CenterCross™ Ultra, CenterCross™ Ultra LV, and/or MultiCross™ devices.

Adverse Events will be coded according to Medical Dictionary for Regulatory Activities (MedDRA). Data from the study will be collected via electronic data capture (EDC). Clinical data will be extracted in the desired format by the BTG Data Management from the EDC on an ongoing basis to support data review activities. An independent monitor will visit the investigational site and review the Electronic Case Report Forms (eCRFs). Data entered in the EDC will be immediately saved to a central database and changes tracked to provide an audit trail.

ELIGIBILITY:
Inclusion Criteria:

* Roxwood CenterCross™, CenterCross™ Ultra, CenterCross™® Ultra LV, MultiCross™ and MicroCross™ 14, 14ES and 18 MicroCatheter device(s) used in first attempts at crossing the stenotic lesion or CTO
* CTO lesion >3 months
* Thrombolysis in myocardial infarction (TIMI) 0 or 1
* Coronary lesion of at least 2.5 millimeter (mm) in diameter
* Native arterial lesions only
* Peripheral lesions no minimum diameter or length
* Adult aged 25 - 80
* Participant understands and has signed the study informed consent form
* Left ventricle ejection fraction >25% (coronary enrollments only)

Exclusion Criteria:

* Endovascular revascularization or surgical revascularization of target lesion within <30 days of procedure
* Prior attempted CTO revascularization (during same procedure)
* Participant unable to give informed consent
* Elevated creatine kinase-muscle/brain (CK-MB) or Troponin levels at baseline
* Participant is known or suspected to be unable to tolerate the contrast agent even with pre-treatment
* CTO is located in aorto-ostial location, saphenous vein graft (SVG), or in-stent
* Appearance of a fresh thrombus or intraluminal filling defects
* Intolerance to Aspirin and/or the inability to tolerate a second antiplatelet agent (Clopidogrel, Prasugrel, Ticagrelor)
* Severe renal insufficiency with estimated glomerular filtration rate (eGFR) <30 milliliters/ minute (mL/min)/1.72 meter squared (m^2)
* Congestive heart failure [New York Heart Association (NYHA) Class III\IV] CSA Class IV
* Life expectancy <6 months due to other illnesses
* Vascular graft
* Women with a positive pregnancy test
* Nitinol or nickel allergy
* Transplanted heart
* Acute or unstable medical disorder/disease that may cause a risk to participant, including:

  * Recent myocardial infarction (MI) <30 days
  * Significant anemia (for example, hemoglobin <8.0 milligram/deciliter (mg/dL)
  * Recent major cerebrovascular event (history of stroke or transient ischemic attack [TIA] within <30 days)
  * Severe uncontrolled systemic hypertension (for example, >180/100 millimeter of mercury [mmHg])
  * Unstable angina requiring emergent percutaneous trans-luminal coronary angioplasty (PTCA) or coronary artery bypass graft (CABG) <30 days

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with chronic total occlusions or stenotic lesions will be screened. The chronic lesions must have occluded the arteries for at least 3 months or longer to be included in this study. Participants undergoing percutaneous revascularization of the native coronary or peripheral vessel where a Roxwood CenterCross™, CenterCross™ Ultra, CenterCross™ Ultra LV, MultiCross™, and MicroCross™ 14, 14ES and 18 MicroCatheter device may be utilized in an attempt at crossing a stenotic lesion or CTO. Up to 12 investigational sites in the United States will participate in this study.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-10-31 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with a Successful Index Procedure by Roxwood Medical Device(s) | Index Procedure (Day 0) to 24 hours Post Procedure
  The number of participants who are successfully treated for an index procedure by Roxwood Medical device(s) to facilitate a guidewire successfully penetrating the proximal cap of a stenotic lesion or CTO and, the infusion of saline and contrast agents, as confirmed by angiography will be measured.
Number of Participants Without an Index Procedure Related Safety Incident Related to the Roxwood Medical Device | Index Procedure (Day 0) to 24 hours Post Procedure
  An index procedure safety incident related to the Roxwood Medical Device is defined as a distal embolization, major perforation or dissection in need of emergent surgical intervention as confirmed by angiography, and bleeding (change from baseline hemoglobin >3 grams/deciliter [g/dL]).

SECONDARY OUTCOMES:
Number of Participants Without an Incidence of a Major Adverse Cardiac Events (MACE) and Urgent Target Vessel Revascularization (TVR) Related to the Roxwood Medical Device | Index Procedure (Day 0) up to Day 30 Post Procedure
  The number of participants without an incidence of a MACE and TVR including, coronary artery bypass graft (CABG) and limb salvage related to the Roxwood Medical device will be measured.
Number of Participants Without Contrast Induced Renal Failure | Baseline up to 24 hours post procedure
  Contrast induced renal failure is defined as a 25% increase in creatinine from Baseline through 24 hours post-procedure.
Time From the Roxwood Medical Device Insertion to Penetration of the Stenotic Lesion or Proximal Cap | Day 0
  The penetration time at Day 0 will be calculated as the time from insertion of the Roxwood Medical device(s) until stenotic lesion or CTO proximal cap penetration.
Time From the Roxwood Medical Device to Cross the True Lumen Distally | Day 0
  The cross time at Day 0 will be calculated as the time from insertion of the Roxwood Medical device(s) until cross the true lumen distally.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Davis, MD, Principal Investigator — Ascension St John
Locations (11):
- United States (11):
  - Dignity Health d/b/a St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Cardiovascular Research of North Florida LLC, Gainesville, Florida
  - St. Mary Medical Center, Inc., Hobart, Indiana
  - MedStar Health Research Institute, Inc., Hyattsville, Maryland
  - Ascension St. John Hospital, Detroit, Michigan
  - McLaren Healthcare Corporation, Flint, Michigan
  - McLaren Healthcare Corporation, Grand Blanc, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Columbia University, New York, New York
  - WellSpan Health Corporation, York, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island